CLINICAL TRIAL: NCT04426409
Title: Effect of Nasal Ointment on Epistaxis of Nasotracheal Intubation in Children: A Randomized Controlled Trial
Brief Title: Nasal Ointment on Epistaxis of Nasotracheal Intubation in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, yun jeong chae, Professor, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AJIRB-MED-INT-19-508
Record Dates: First submitted 2020-06-08; First posted 2020-06-11 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Epistaxis; Intubation
MeSH Terms: conditions — Epistaxis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention)
- ointment group (Experimental): Ointment group should apply a nasal ointment to both noses using a cotton swab the night before surgery and the morning of surgery.
  Interventions: Drug: tarivid ointment

INTERVENTIONS:
Drug: tarivid ointment — Vaseline ointment is applied to both noses.
  Arms: ointment group

SUMMARY:
Nasotracheal intubation is one of the anesthetic procedures required for oral surgery. It allows the surgeon easier access to the surgical site than the orthotracheal intubation. Therefore, nosotracheal intubation is commonly used for general anesthesia for oral and maxillofacial surgery and dental treatment. However, nasotracheal intubation can damage the nasal mucosa in the course of the tube passing through the nostrils, causing epistaxis which is reported as the most common side effect.

In order to reduce these side effects, heating of the tube and use of a tube lubricant immediately before intubation have been recommended in children. However, research on whether the dry state of the mucosa itself contributes to the development of epistaxis is limited. A study in adults reported that pretreatment of the ointment on the mucosa reduced the damage to the mucosa. However, its effect on the incidence of epistaxis in children has not been studied.

The purpose of this study is to investigate the effects of pretreatment of nasal ointment on epistaxis of nasotracheal intubation in children.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical statue I or II
* Patients scheduled to undergo surgery under nasotracheal intubation

Exclusion Criteria:

* expected difficult intubation based on history, physical examination, weight.
* bleeding tendency
* upper respiratory infection within the previous 14 days

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 108 (Actual)
Dates: Start 2020-07-08 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
incidence of epistaxis | immediate after intubation
  percentage of the development of epistaxis after nasotracheal intubation
incidence of epistaxis | immediate after extubation
  percentage of the development of epistaxis after nasotracheal intubation

SECONDARY OUTCOMES:
severity of epistaxis | immediate after intubation
  score based on severity of epistaxis will be recorded.
  1: no epistaxis, 2: mild; blood on tube 3. moderate: blood pooling on pharynx 4. severe: interfere intubation by blood
severity of epistaxis | immediate after extubation
  score based on severity of epistaxis will be recorded.
  1: no epistaxis, 2: mild; blood on tube 3. moderate: blood pooling on pharynx 4. severe: interfere intubation by blood
Navigability | immediate after intubation
  score based on easiness of navigation during intubation
  1. No resistance 2. Pass with some resistance(1try, mild) 3. Pass with some resistance (>=2) 4. Failed to pass (Try to another nose) 5. Failed to pass both nostril (use more smaller tube)

CONTACTS AND LOCATIONS:
Locations (1):
- Ajou University School of Medicine, Suwon, Gyeonggi-do, South Korea